CLINICAL TRIAL: NCT02552004
Title: Assessment of the Intraoperative Probe-based Confocal Laser Endomicroscopy in Digestive and Endocrine Surgery - a Pilot Study
Brief Title: Assessment of Intraoperative Probe-based Confocal Laser Endomicroscopy in Digestive and Endocrine Surgery: a Pilot Study
Acronym: Pilot pCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-001
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: All Surgical Conditions Usually Necessitating Frozen Section; Malignant Tumor; Inflammatory Disease; Benign Tumor
Keywords: pCLE; Digestive surgery; Endocrine surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pCLE (Experimental): Patients subject to endocrine or digestive surgery will have intraoperative pCLE examination. The installation and surgical opening will be performed according to standard protocols. The contrast agent, fluorescein, will be injected intravenously to allow tissue visualization with pCLE. During the surgery, the surgeon will perform the pCLE examination, to obtain and record video sequences of in situ structures. Frozen sections will be obtained on the same samples and will further guide the surgical decision-making.
  Interventions: Device: pCLE; Drug: IV fluorescein administration

INTERVENTIONS:
Device: pCLE — Histological examination by pCLE technique preceding the frozen section
Drug: IV fluorescein administration — IV Fluorescein (fluorescent contrast agent) administration

SUMMARY:
Intraoperative histological examination is a fundamental tool in surgery. Probe-based Confocal Laser Endomicroscopy (pCLE) is a new imaging technique which enables real-time, microscope-resolution imaging, currently used in endoscopy. This pilot study aims to evaluate pCLE in surgical setting. The objective is the depiction of histological rendering of normal and pathological tissues through pCLE. Feasibility of real-time diagnosis will also be assessed. All surgical conditions usually necessitating frozen section will be investigated. A total of 30 patients, with various pathology of the thyroid / parathyroid, stomach, esophagus, pancreas, adrenal, colon / small intestine, liver will be included. Diagnostic criteria will be defined by a surgeon - pathologist team and further validated by retrospective analysis of the video sequences in comparison to conventional histology slides. The data will be used to create an image bank of reference optical biopsy images. The study will allow to point out the surgical conditions in which pCLE is the most effective and reliable and could eventually replace the frozen section technique.

DETAILED DESCRIPTION:
Intraoperative histological examination is a fundamental tool for cancer surgery (extent of surgery, resection margins, sentinel lymph node) and necessary in other circumstances like redo surgery or endocrine surgery. Using conventional frozen section technique results in the prolongation of operating time of about 40 minutes.

Probe-based Confocal Laser Endomicroscopy (pCLE) is a new imaging technique which enables real-time, microscope-resolution imaging. Specifically, after intravenous injection of a fluorescent contrast agent - in this study fluorescein will be used, the pCLE system provides video sequences of the tissue, using a confocal microscope integrated in a miniprobe and a low power laser as the illumination source (Cellvizio®, Mauna Kea Technologies, Paris, France).

The pCLE is currently used in endoscopy, mainly for the follow-up of Barrett's esophagus, colorectal polyps and strictures of the bile and pancreatic ducts, but also in urology. The pCLE has never been tested in open or video-assisted surgery settings. Sterilizable probes exist and are certified for use via an endoscope in France (UHD CystoFlexTM, AQ-FLEX 19TM Mauna Kea Technologies, Paris, France). A probe (CelioFlex UHDTM) is currently being developed for use in laparoscopic surgery setting.

This pilot study aims to evaluate pCLE in surgical setting. Each anatomical structure corresponds to a specific tissue architecture, which is today known through standard histological examination. Conventional histology implies alteration of the tissue architecture, with ablation of blood supply, sampling and technical treatment of the samples (fixation, cutting, staining). The pCLE enables to bypass this process and allows obtaining images of the microscopic structure in vivo, without cell damage and without interruption of the blood and lymphatic circulation. The obtained video sequences reflect the microscopic architecture, in a form which is to date, neither mapped nor exploited for deep organs. The potential of this technique was demonstrated in intraabdominal organs only in the animal model, with very encouraging results as the sensitivity and specificity of pCLE were superior to standard histological examination.

The primary objective is the depiction of histological rendering of normal and pathological tissues through pCLE. Feasibility of real-time diagnosis will also be assessed. All surgical conditions usually necessitating frozen section will be investigated. A total of 30 patients, with various pathology of the thyroid / parathyroid, stomach, esophagus, pancreas, adrenal, colon / small intestine, liver will be included.

The installation and surgical opening will be performed according to standard protocols. A contrast agent, fluorescein, will be injected intravenously to allow tissue visualization with the pCLE. During the surgery, the surgeon will perform the pCLE examination, to obtain and record video sequences of in situ structures. Frozen sections will be obtained on the same samples and will further guide the surgical decision-making.

Diagnostic criteria will be defined by a surgeon - pathologist team and further validated by retrospective analysis of the sequences in comparison to conventional histology slides. The data will be used to create an image bank of reference optical biopsy images.

The study will allow to point out the surgical conditions in which pCLE is the most effective and reliable and could eventually replace the frozen section technique.

A second study, in comparative prospective settings, could further be focused only on the promising conditions in order to evaluate diagnosis accuracy on a statistical basis.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old
* Patient candidate to digestive or endocrine surgery in whom the surgeon deems necessary intraoperative frozen section
* Patient able to understand the study and to provide informed consent
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient unable to provide informed consent
* Patient with known or suspected allergy to fluorescein
* Patient who had a previous life-threatening reaction during an angiography
* Patient with a history of multiple and severe allergic reactions to medications
* Patient taking a beta-blocker treatment
* Patient with comorbidity considered by the investigator, as incompatible with the procedures of the study
* Patient pregnant or breastfeeding
* Patient in exclusion period (determined by a previous study or in progress)
* Patient having forfeited their freedom of an administrative or legal obligation
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis accuracy of intraoperative imaging with pCLE technique | During surgery
  The diagnosis proposed by the surgeon / investigator in intraoperative setting on the basis of video sequences of pCLE will be compared to frozen section.

SECONDARY OUTCOMES:
Diagnosis accuracy of pCLE imaging, retrospectively using the newly described diagnosis criteria | One year
  The diagnosis proposed by the surgeon / investigator after retrospective review of the intraoperative video sequences of pCLE based on the newly described diagnosis criteria will be compared to frozen section and conventional histology.
pCLE video sequences interpretation learning curve | One year
  Comparison of the surgeon's ability to obtain intraoperative diagnosis relative to that of the pathologist in the same circumstances.
Time needed for pCLE imaging procedure | During surgery
  Evaluation of the time required for the practice of pCLE and comparison to the time required for frozen section.
Specific morbidity and mortality rate | One month after surgery
  Morbidity rate / mortality specific to the pCLE imaging procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Ignat, MD, PhD, Principal Investigator — Service de chirurgie digestive et endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de chirurgie digestive et endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Background] Wallace MB, Fockens P. Probe-based confocal laser endomicroscopy. Gastroenterology. 2009 May;136(5):1509-13. doi: 10.1053/j.gastro.2009.03.034. Epub 2009 Mar 28. No abstract available. PMID 19328799
- [Background] Ignat M, Aprahamian M, Lindner V, Altmeyer A, Perretta S, Dallemagne B, Mutter D, Marescaux J. Feasibility and reliability of pancreatic cancer staging using fiberoptic confocal fluorescence microscopy in rats. Gastroenterology. 2009 Nov;137(5):1584-92.e1. doi: 10.1053/j.gastro.2009.07.045. Epub 2009 Jul 24. PMID 19632230
- [Background] Kwan AS, Barry C, McAllister IL, Constable I. Fluorescein angiography and adverse drug reactions revisited: the Lions Eye experience. Clin Exp Ophthalmol. 2006 Jan-Feb;34(1):33-8. doi: 10.1111/j.1442-9071.2006.01136.x. PMID 16451256
- [Result] Ignat M, Lindner V, Vix M, Marescaux J, Mutter D. Intraoperative Probe-Based Confocal Endomicroscopy to Histologically Differentiate Thyroid From Parathyroid Tissue Before Resection. Surg Innov. 2019 Apr;26(2):141-148. doi: 10.1177/1553350618814078. Epub 2018 Nov 23. PMID 30466375